CLINICAL TRIAL: NCT06478199
Title: PLR and NLR as Predictor Factors for Semen Abnormality
Status: Active, not recruiting | Type: Observational
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Elsayed Abdelhalim Elsayed, assistant lecturer of urology, Kafrelsheikh University
Other Study IDs: semen paramaters
Record Dates: First submitted 2024-06-24; First posted 2024-06-27 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Fertility Issues
MeSH Terms: conditions — Infertility | interventions — Semen Analysis; Blood Cell Count

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A :normal semen
  Interventions: Diagnostic Test: semen analysis
- Group B : abnormal semen
  Interventions: Diagnostic Test: semen analysis

INTERVENTIONS:
Diagnostic Test: semen analysis — lab invesigation
  Other Names: cbc

SUMMARY:
The aim of this study was to evaluate the relationship of seminal parameters with the neutrophil-to-lymphocyte ratio (NLR) and the platelet-to-lymphocyte ratio (PLR), which are inflammatory markers, in men with an abnormal semen analysis and men with normozoospermia.

ELIGIBILITY:
Inclusion Criteria:

* adult above 18 years primary not do varicocelectomy

Exclusion Criteria:

* young secondry infertility recurrent varicocele

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient correlat to inclusion criteria
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Laboratory result | 1 day
  cbc and semen analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided